CLINICAL TRIAL: NCT03246230
Title: Systems Biology to Identify Biomarkers of Neonatal Vaccine Immunogenicity
Acronym: EPIC-HIPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other); University of British Columbia (Other); Institute for Medical Research, Papua New Guinea (Unknown); The University of Western Australia (Other)
Responsible Party: Principal Investigator, Ofer Levy, Staff Physician, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-P00024239
Record Dates: First submitted 2017-08-04; First posted 2017-08-11 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Newborn Vaccine Immunogenicity
Keywords: newborn vaccine responses
MeSH Terms: interventions — Hepatitis B Vaccines

STUDY DESIGN:
Intervention Model Description: Newborn infants will have delayed immunization, with catch-up immunization at day of life 7 (DOL7), or immunization at birth with hepatitis B vaccine (HBV), Bacille Calmette-Guérin (BCG) or (HBV +BCG). All participants will have peripheral blood collected at birth (DOL0) and each group will be divided into sub-groups with follow-up peripheral blood collection at DOL1, DOL3, or DOL7.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NO VACCINES AT BIRTH (No Intervention): These will be newborns who will not receive any vaccines at birth and will have delayed immunization with catch-up (i.e., HBV, BCG and polio vaccine) by Day of Life 7.
- HBV VACCINE AT BIRTH (Other): Participants in this arm will receive licensed hepatitis B vaccine (HBV) at birth (Day of Life (DOL)-0) with catch up immunization (i.e., BCG and polio vaccine) at DOL-1, -3, or -7.
  Interventions: Biological: Hepatitis B vaccine (HBV)
- BCG VACCINE AT BIRTH (Other): Participants in this arm will receive licensed Bacillus Calmette-Guérin (BCG) vaccine at birth (Day of Life(DOL)-0) with catch up immunization (i.e., HBV and polio vaccine) at DOL-1, -3 or- 7.
  Interventions: Biological: Bacillus Calmette-Guérin (BCG)
- (HBV + BCG) VACCINES AT BIRTH (Other): Participants in this arm will receive licensed hepatitis B vaccine (HBV) and licensed Bacillus Calmette-Guérin (BCG) vaccine at birth (Day of Life (DOL- 0) with catch up immunization (i.e., polio vaccine) at DOL-1, -3, or -7.
  Interventions: Biological: Hepatitis B vaccine (HBV); Biological: Bacillus Calmette-Guérin (BCG)

INTERVENTIONS:
Biological: Hepatitis B vaccine (HBV) — Licensed pediatric HBV vaccine will be administered at birth (Day of Life 0) or delayed to Day of Life 7.
  Arms: (HBV + BCG) VACCINES AT BIRTH; HBV VACCINE AT BIRTH
Biological: Bacillus Calmette-Guérin (BCG) — Licensed BCG vaccine will be administered at birth (Day of Life 0) or delayed to Day of Life 7.
  Arms: (HBV + BCG) VACCINES AT BIRTH; BCG VACCINE AT BIRTH

SUMMARY:
Infection is the most common cause of death in early life, especially for newborns and can be reduced by immunization but insufficient knowledge of how vaccines protect the very young limits their optimal use. To gain insight into how vaccines induce protection of the most vulnerable, this National Institutes of Health (NIH)/National Institute of Allergy & Infectious Diseases (NIAID)-funded Human Immunology Project Consortium (HIPC) study, based at Boston Children's Hospital and conducted by the Expanded Program on Immunization Consortium (EPIC), employs two novel approaches studying newborn responses to hepatitis B vaccine (HBV): (a) systems biology that uses technologies which comprehensively measure global changes in molecules such as transcriptomics (RNA) and proteomics (proteins), as well as cell composition of the blood and (b) use of human newborn blood components, collected prior to immunization, to model vaccine responses in vitro (outside the body). Characterizing vaccine-induced molecular patterns ("signatures") that correspond to vaccine-mediated protection will accelerate development and optimization of vaccines against early life infections of major global health importance.

DETAILED DESCRIPTION:
While the greatest number of vaccines is administered to the very young, vaccine preventable infections remain a major cause of morbidity and mortality, especially for the newborn. To improve vaccine-mediated protection early in life, the investigators will identify biomarkers that predict protective efficacy and garner insight into the underlying mechanisms of vaccine-mediated protection. Systems biology approaches ("OMICs") applied to vaccinology, i.e., systems vaccinology, has revolutionized the field with an unbiased identification of pathways relevant to vaccine-induced immune responses. However, thus far systems vaccinology has focused primarily on adults, with few studies conducted in children and infants, and none in newborns. This study will bridge this gap by conducting a comprehensive systems vaccinology study in newborns. Specifically, the investigators will determine the molecular pathways that are associated with successful neonatal immunization with hepatitis B virus vaccine (HBV). HBV is the ideal model because i) it is highly (>90%) effective; ii) it has a well-established correlate of protection (CoP; anti-hepatitis surface antigen antibody (anti-HBs)); iii) there is substantial variation in anti-HBs titers and quantifiable inter-subject variability is essential for systems biological approaches; iv) it is highly relevant as HBV is given at birth in the U.S. and most developing countries; v) it is amenable to in vivo manipulation with another regularly administered neonatal vaccine, Bacille Calmette-Guérin (BCG), which will greatly enhance detection of relevant signatures. As complex networks of functional interactions among genes and proteins drive the response to immunization, the investigators will integrate transcriptomic, proteomic and immune phenotyping approaches. Importantly, the investigators have successfully adapted these experimental platforms to be fully operational within the small blood volumes obtainable in newborns. The investigators have also developed in vitro systems amenable to experimental manipulation on the cellular and molecular level to identify cause-effect relationships. Pilot data prove feasibility of collecting the relevant high-quality samples according to stringent standard operating procedures, processing them and delivering cogent OMIC data suggesting vaccine-specific 'signatures' in the human newborn. This HIPC will identify biomarkers of neonatal HBV immunogenicity by pursuing the following Overall Specific Aims:

* Aim 1. Characterize pre-vaccine OMIC and immune signatures in vivo that predict immunogenicity of HBV in human newborns. In adult systems vaccinology studies, baseline immune status of vaccine recipients predicted vaccine immunogenicity at least as well or even better than changes induced by the vaccine. For Aim 1 the investigators will determine the pre-vaccine (Day 0) characteristics of whole blood gene expression, plasma proteome as well as the composition of the white blood cell compartment and their functional status in correlation with the HBV-induced neonatal antibody response.
* Aim 2. Characterize the post-vaccine impact of HBV on OMIC and immune signatures in vivo that predict immunogenicity of HBV in human newborns. In adults, analysis of vaccine-induced signatures (i.e. post-vaccine) has provided new insights for several vaccines, including HBV. The investigators will for the first time apply this approach to newborns and expand it by manipulating the neonatal response to HBV in vivo by co-administering BCG, as it substantially changes immunogenicity of HBV thereby testing cause-effect relationships in vivo. For Aim 2 the investigators will characterize whole blood gene expression and the plasma and leukocyte proteome as well as white blood cell composition and functional status at Days 1, -3 and -7 postvaccine contrasting infants that received nothing (delayed vaccines to 7 days of age), HBV, BCG or (HBV + BCG) at birth and correlate this with anti-HBs titers.
* Aim 3. Interrogate functional correlations identified in silico via novel human in vitro platforms that accurately model age-specific vaccine responses and are amenable to a wide range of experimental manipulation allowing mechanistic cause-effect relationships to be probed on the molecular level.

Overall, these integrated studies will identify vaccine-induced molecular pathways correlating with protective immune responses in newborns and will generate and test new mechanistic hypotheses regarding vaccine action in vivo and in vitro. This study will ultimately inform, accelerate and optimize early life immunization resulting in major public health benefit.

ELIGIBILITY:
Inclusion Criteria:

* <24 hours of age
* >37 weeks gestational age
* HIV unexposed
* Healthy (no malformations, normal temperature range and vital signs for age)

Exclusion Criteria:

* Premature (<37 weeks gestational age)
* Hepatitis B antigen-positive mother
* HIV-positive or HIV-exposed
* Febrile, unstable vital signs

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 911 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
Molecular signature correlating with anti-hepatitis B vaccine antibody response | 1 month of age
  We will employ bioinformatics to define molecular signatures correlating with anti-HBV responses

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Levy, MD, PhD, Principal Investigator — Boston Children's Hospital; Tobias R Kollmann, MD, PhD, Study Director — The University of Western Australia; Beate Kampmann, MD, PhD, Study Chair — Medical Research Council (MRC) Gambia
Locations (2):
- Institute for Medical Research, Goroka, Eastern Highlands Province, Papua New Guinea
- Medical Research Council Unit, The Gambia, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amenyogbe N, Levy O, Kollmann TR. Systems vaccinology: a promise for the young and the poor. Philos Trans R Soc Lond B Biol Sci. 2015 Jun 19;370(1671):20140340. doi: 10.1098/rstb.2014.0340. PMID 25964462
- [Background] Lee AH, Shannon CP, Amenyogbe N, Bennike TB, Diray-Arce J, Idoko OT, Gill EE, Ben-Othman R, Pomat WS, van Haren SD, Cao KL, Cox M, Darboe A, Falsafi R, Ferrari D, Harbeson DJ, He D, Bing C, Hinshaw SJ, Ndure J, Njie-Jobe J, Pettengill MA, Richmond PC, Ford R, Saleu G, Masiria G, Matlam JP, Kirarock W, Roberts E, Malek M, Sanchez-Schmitz G, Singh A, Angelidou A, Smolen KK; EPIC Consortium; Brinkman RR, Ozonoff A, Hancock REW, van den Biggelaar AHJ, Steen H, Tebbutt SJ, Kampmann B, Levy O, Kollmann TR. Dynamic molecular changes during the first week of human life follow a robust developmental trajectory. Nat Commun. 2019 Mar 12;10(1):1092. doi: 10.1038/s41467-019-08794-x. PMID 30862783
- [Derived] Montante S, Ben-Othman R, Amenyogbe N, Angelidou A, van den Biggelaar A, Cai B, Chen Y, Darboe A, Diray-Arce J, Ford R, Idoko O, Lee A, Lo M, McEnaney K, Malek M, Martino D, Masiria G, Odumade OA, Pomat W, Shannon C, Smolen K, Consortium TE, Ozonoff A, Richmond P, Tebbutt S, Levy O, Kampmann B, Brinkman R, Kollmann T. Breastfeeding and Neonatal Age Influence Neutrophil-Driven Ontogeny of Blood Cell Populations in the First Week of Human Life. J Immunol Res. 2024 Jul 23;2024:1117796. doi: 10.1155/2024/1117796. eCollection 2024. PMID 39081632
- [Derived] Idoko OT, Smolen KK, Wariri O, Imam A, Shannon CP, Dibassey T, Diray-Arce J, Darboe A, Strandmark J, Ben-Othman R, Odumade OA, McEnaney K, Amenyogbe N, Pomat WS, van Haren S, Sanchez-Schmitz G, Brinkman RR, Steen H, Hancock REW, Tebbutt SJ, Richmond PC, van den Biggelaar AHJ, Kollmann TR, Levy O, Ozonoff A, Kampmann B. Clinical Protocol for a Longitudinal Cohort Study Employing Systems Biology to Identify Markers of Vaccine Immunogenicity in Newborn Infants in The Gambia and Papua New Guinea. Front Pediatr. 2020 Apr 30;8:197. doi: 10.3389/fped.2020.00197. eCollection 2020. PMID 32426309
- See also: Human Immunology Project Consortium/National Institute of Allergy & Infectious Diseases — https://www.niaid.nih.gov/research/human-immunology-project-consortium
- See also: Precision Vaccines Program, Boston Children's Hospital — https://www.childrenshospital.org/research/departments/pediatrics-research/precision-vaccines-program
- See also: Data, Tools & Resources related to NIH/NIAID Human Immunology Project Consortium — https://immunespace.org